CLINICAL TRIAL: NCT03294317
Title: Imagining Study of Lead Implant for His Bundle Pacing
Brief Title: Imaging Study of Lead Implant for His Bundle Pacing
Acronym: (IMAGE-HBP)
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: IMAGE-HBP
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Results first posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Cardiac Pacemaker, Artificial
Keywords: His bundle pacing; Pacemaker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- His Bundle Pacing: Patient will be implanted per indications for single or dual chamber pacemaker. Lead for His bundle pacing will be implanted.
  Interventions: Device: His bundle pacing

INTERVENTIONS:
Device: His bundle pacing — Medtronic SelectSecure SureScan MRI model 3830 lead

SUMMARY:
The purpose of this research study is to assess the implant success proportion of the Medtronic SelectSecure MRI SureScan Model 3830 pacing lead at the bundle of His for His bundle pacing.

DETAILED DESCRIPTION:
The study will evaluate implant lead electrical measurements and changes over time, estimate the correlation between lead location and selective vs non-selective His bundle pacing, and estimate the correlation between long-term lead performance and implant characteristics. Data from the study may be used to standardize the implant workflow to help improve the ease and predictability of His bundle pacing implants.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a Class I or II indication for implantation of an implantable pacemaker
* Subject (or legally authorized representative) has signed and dated the study-specific Consent Form
* Subject is 18 years of age or older, or is of legal age to give informed consent per local and national law
* Subject is expected to remain available for follow-up visits

Exclusion Criteria:

* Subject is contraindicated for Cardiac CT
* Subject has an existing or prior pacemaker, ICD or CRT device implant
* Subject is intended to receive an implant of a LV lead or CRT device
* Subject life expectancy is less than 1 year
* Pregnant women or breastfeeding women, or women of child bearing potential and who are not on a reliable form of birth regulation method or abstinence
* Subjects with exclusion criteria required by local law (e.g. age or other)
* Subject with a medical condition that precludes the patient from participation in the opinion of the investigator
* Subject is enrolled in a concurrent study that may confound the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bradycardia patients, AV Block patients, Sinus Node Dysfunction patients
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2020-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pugazhendhi Vijayaraman, MD, Principal Investigator — Geisinger Wyoming Valley Medical Center
Locations (3):
- United States (3):
  - Indiana University - Krannert Institute of Cardiology, Indianapolis, Indiana
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Virginia Commonwealth University Health System, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vijayaraman P, Dandamudi G, Subzposh FA, Shepard RK, Kalahasty G, Padala SK, Strobel JS, Bauch TD, Ellenbogen KA, Bergemann T, Hughes L, Harris ML, Fagan DH, Yang Z, Koneru JN; IMAGE-HBP Investigators. Imaging-Based Localization of His Bundle Pacing Electrodes: Results From the Prospective IMAGE-HBP Study. JACC Clin Electrophysiol. 2021 Jan;7(1):73-84. doi: 10.1016/j.jacep.2020.07.026. Epub 2020 Sep 30. PMID 33478715

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 subjects signed consent. Per the protocol , a subject is considered enrolled in the study upon signing and dating the informed consent. Of the 70 who signed informed consent, 69 were considered "enrolled" per the protocol. 1 was "screen failure", i.e they signed informed consent, but ended up failing inclusion/exclusion
Pre-assignment Details: Of the 70 subjects who signed informed consent, 1 failed inclusion/exclusion criteria and was exited from the study and left us with 69 subjects. 8 of the 69 subjects were "Implant Attempted" i.e they failed HB lead implant and was exited from the study. 61 subjects had the lead placed at the His-bundle and for various reasons, such as lost to follow-up, physician decision, subject withdrew, received CRT 11 of the subjects were exited leaving us with 50 subjects who completed the study.
Period: Overall Study
Arm/Group | His Bundle Pacing
Started | 70
Implanted With Lead at HIS Bundle | 61
Subjects With Available CT | 51
Completed | 50
Not Completed | 20
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 1
Not completed — Did not meet inclusion/exclusion criteria | 1
Not completed — Failed HB lead implant | 8
Not completed — Received CRT instead | 1
Not completed — Exited after lead revision | 2

BASELINE CHARACTERISTICS:
Population: Baseline demographics and medical history were summarized for all subjects with an implant attempt in the study.
Arm/Group | His Bundle Pacing
Number analyzed (Participants) | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Implant Success
Description: To determine the proportion implant successes from all subjects who undergo an implant attempt of a lead at the bundle of His for His bundle pacing. Implant success will be defined as the presence of a H wave on the implanted lead EGM and a His-bundle pacing capture threshold equal to or less than 2.5V at 1.0ms.
Time Frame: Day of implant
Population: The primary objective is to assess the implant success proportion of the Medtronic Model 3830 pacing lead at the bundle of His for His Bundle Pacing. The observed implant success proportion was calculated as follows:
  Implant Success Proportion= ( # Subjects with implant success)/( # Subjects with implant attempt) The observed implant success proportion was 75.36% and the 95% confidence interval is 64.04% - 84.01%.
Measure: Number (95% Confidence Interval); unit: % of subjects with successful implant
Arm/Group | His Bundle Pacing
Number analyzed (Participants) | 69
% of subjects with successful implant | 75.36 [64.04 to 84.01]

2. Secondary Outcome: Association Between the Lead Position and Selective vs. Nonselective HBP Occurrence at Implant
Description: Relationship between lead position (anterior septum, mid septum, posterior septum) and His-bundle pacing selectivity (selective vs. non-selective)
Time Frame: Day of implant
Population: The lead position is analyzed using two variables. The first variable is whether the lead tip is on the atrial or ventricular side of the TV annulus. The second variable is whether the lead tip is above or below the CS line, on the atrial side, or the RV line, on the ventricular side of the TV. The relationship between lead position was assessed using a logistic regression where the dependent variable was HB pacing type and the independent variables were the two lead position variables.
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | His Bundle Pacing
Number analyzed (Participants) | 51
odds ratio
  Atrial/Ventricular side of TV annulus | 1.27 [0.24 to 6.58]
  Above/Below side of CS/RV line | 0.57 [0.14 to 2.29]

3. Secondary Outcome: Changes in His-bundle Pacing Capture Thresholds Over Time
Description: The change in the His-bundle pacing capture threshold from implant to 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: volts
Arm/Group | His Bundle Pacing
Number analyzed (Participants) | 46
volts | 1.82 (1.03)

4. Secondary Outcome: Changes in Impedance Over Time
Description: To evaluate impedance from implant to 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | His Bundle Pacing
Number analyzed (Participants) | 47
ohms | 429.72 (79.29)

5. Secondary Outcome: Changes in R-wave Amplitude Over Time
Description: To evaluate R-wave amplitude from implant to 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | His Bundle Pacing
Number analyzed (Participants) | 34
millivolts | 4.10 (2.15)

6. Secondary Outcome: Changes in QRS Duration Over Time
Description: Intrinsic QRS duration measured prior to implant procedure and compared to measurements during follow-up
Time Frame: 12 months
Population: The QRS duration measurements evaluated include both intrinsic, paced QRS duration during pacing threshold testing, and paced QRS duration at final programming. Longitudinal analysis was conducted to estimate differences in QRS duration measurements from implant to subsequent follow-up visits using a mixed effects model.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | His Bundle Pacing
Number analyzed (Participants) | 47
milliseconds | 105.00 (32.05)

7. Secondary Outcome: Association Between Lead Location and Long-term Lead Electrical Performance
Description: To assess the association between lead location and long-term lead electrical performance defined by the His-bundle pacing capture threshold at 12 months post-implant.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Regression coefficient
Arm/Group | His Bundle Pacing
Number analyzed (Participants) | 45
Regression coefficient
  Atrial/Ventricular side of TV annulus | 0.070681015 [-0.587845 to 0.729207]
  Above/Below side of CS/RV line | 0.106436807 [-0.439328 to 0.652202]

8. Secondary Outcome: Correlation Between His-bundle Pacing Capture Threshold at Implant and Long-term Lead Electrical Performance
Description: To assess the correlation between His-bundle pacing capture threshold at implant and long-term lead electrical performance defined by the His-bundle pacing capture threshold at 12 months post-implant.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Regression coefficient
Arm/Group | His Bundle Pacing
Number analyzed (Participants) | 45
Regression coefficient | 0.308729841 [0.008103 to 0.609357]

9. Secondary Outcome: Correlation Between Paced QRS Duration at Implant and Long-term Lead Electrical Performance
Description: To assess the correlation between paced QRS duration at implant and long-term lead electrical performance defined by the His-bundle pacing capture threshold at 12 months post-implant.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Regression coefficient
Arm/Group | His Bundle Pacing
Number analyzed (Participants) | 45
Regression coefficient | -0.001329355 [-0.012422 to 0.009763]

10. Secondary Outcome: Complications Related to the Procedure or the Lead for His Bundle Pacing
Description: Adverse events that are complications related to the procedure or the lead for His bundle pacing will be summarized
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | His Bundle Pacing
Number analyzed (Participants) | 69
participants | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 12 months
Arm/Group | His Bundle Pacing
All-Cause Mortality (participants affected / at risk) | 0/69
Serious Adverse Events (participants affected / at risk) | 3/69
Other Adverse Events (participants affected / at risk) | 3/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | His Bundle Pacing (N=69)
Device capturing issue (Cardiac disorders) | 1 (1)
Device pacing issue (Cardiac disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | His Bundle Pacing (N=69)
Device pacing issue (Cardiac disorders) | 1 (1)
Bundle branch block right (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator and Participating Institution shall submit any contemplated publication or presentation of this study to Medtronic for review at least 60 days prior to submission, If notified by Medtronic within such 60- day period that such publication or presentation contains Confidential Information, Investigator and Participating Institution each agree to delete Confidential Information, other than Study results, prior to any publication or presentation.

DOCUMENTS (3):
  • Study Protocol (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT03294317/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT03294317/SAP_001.pdf
  • Informed Consent Form (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT03294317/ICF_002.pdf